CLINICAL TRIAL: NCT07134270
Title: Association Between Digestive MDRO Carriage and Infection Risk in Hospitalized Patients: A Single-Center Prospective Analysis
Brief Title: Infection Risk Associated With Digestive MDRO Carriage in Hospitalized Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Valeriu Gheorghita (Other)
Responsible Party: Sponsor-Investigator, Valeriu Gheorghita, Prof. Univ. Dr., Emergency and Clinical Hospital "Dr. Agrippa Ionescu"
Organization: Emergency and Clinical Hospital "Dr. Agrippa Ionescu" (Other)
Other Study IDs: 289334/29.04.2025
Record Dates: First submitted 2025-07-16; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Multi Drug Resistant Organisms
Keywords: MDRO; ESBL; CRE; CRPA; CRAB; VRE; hospital-acquired infections; digestive carriage; antimicrobial resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — rectal swabs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MDRO Carriers: Patients with confirmed digestive (rectal) carriage of multidrug-resistant organisms (MDRO), detected through rectal swab at admission. These include ESBL-producing Enterobacterales, CRE, CRPA, CRAB, and VRE.
  Interventions: Procedure: MDRO Rectal Screening; Other: 30-Day Telephone Follow-Up
- Non-Carriers: Patients with negative screening for MDRO carriage at admission. These individuals serve as the control cohort for assessing infection risk in the absence of digestive colonization at admission.
  Interventions: Procedure: MDRO Rectal Screening; Other: 30-Day Telephone Follow-Up

INTERVENTIONS:
Procedure: MDRO Rectal Screening — Repeated rectal swab collection for screening digestive colonization with multidrug-resistant organisms (MDRO), performed at admission (or within 14 days prior), on day 7, weekly during hospitalization, and at discharge.
Other: 30-Day Telephone Follow-Up — Structured phone interview conducted 30 days post-discharge, using a standardized questionnaire assessing new infections, rehospitalizations, antibiotic use, and self-rated health status.

SUMMARY:
This study aims to evaluate the impact of digestive carriage of multidrug-resistant organisms (MDRO) on the risk of healthcare-associated infections in hospitalized adult patients. Patients will be screened at admission, weekly, and at discharge, with a 30-day post-discharge follow-up. The findings will support infection prevention and control strategies in Romanian hospitals.

DETAILED DESCRIPTION:
This is a prospective, observational cohort study conducted at the Clinical Emergency Hospital "Prof. Dr. Agrippa Ionescu" in Bucharest, Romania. The study aims to assess the epidemiology and clinical impact of digestive colonization with multidrug-resistant organisms (MDRO) in hospitalized adult patients. MDROs of interest include extended-spectrum beta-lactamase-producing Enterobacterales (ESBL), carbapenem-resistant Enterobacterales (CRE), carbapenem-resistant non-fermenting Gram-negative bacilli (Pseudomonas aeruginosa, Acinetobacter baumannii), and vancomycin-resistant Enterococcus spp. (VRE).

Eligible participants are ≥18 years old and admitted to one of the following hospital departments: General Surgery, Internal Medicine, Infectious Diseases, Hematology, Oncology, or Intensive Care Unit (ICU). A minimum of 400 patients will be enrolled and followed during hospitalization and up to 30 days post-discharge.

Upon enrollment, patients will undergo rectal swab screening for MDRO carriage at baseline (within 14 days prior to or at admission), on day 7 of hospitalization, weekly thereafter, and at discharge. Data on comorbidities (including Charlson Comorbidity Index), prior hospitalizations or surgeries, recent antibiotic exposure, and potential epidemiologic risk factors (e.g., travel to endemic areas) will be collected.

The primary objective is to assess the cumulative risk of developing healthcare-associated infections (HAIs) during hospitalization in patients with digestive carriage of MDRO compared to those without. Secondary objectives include:

Estimation of the MDRO carriage prevalence at admission;

Assessment of conversion from negative to positive carriage during hospitalization;

Characterization of clinical and epidemiologic profiles associated with MDRO carriage;

Identification of etiologic patterns and resistance mechanisms.

A structured follow-up by telephone will be conducted 30 days after discharge, including a standardized questionnaire assessing new infections, rehospitalizations, antibiotic use, and perceived health status.

Collected microbiological data may be correlated with molecular characterization (e.g., resistance genes, phylogenetic analysis) through collaboration with the "Cantacuzino" National Institute for Research and Development in Military Medicine.

All procedures comply with the Declaration of Helsinki and GDPR regulations. Participation is voluntary, and patients may withdraw at any time without consequences for their medical care

ELIGIBILITY:
Inclusion Criteria:

* 18 years

Admitted to participating wards

Signed informed consent

Exclusion Criteria:

* withdrawal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) admitted to medical and surgical departments of the Clinical Emergency Hospital "Prof. Dr. Agrippa Ionescu" in Bucharest, Romania, including Internal Medicine, Infectious Diseases, Hematology, Oncology, General Surgery, and Intensive Care Unit. Participants are enrolled consecutively and undergo screening for digestive MDRO carriage during hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of healthcare-associated infections during hospitalization | Up to 30 days after discharge
  Rate of infections in MDRO carriers versus non-carriers.

SECONDARY OUTCOMES:
Prevalence of MDRO Digestive Carriage at Admission | Within 48 hours of hospital admission
  Proportion of participants testing positive for digestive colonization with multidrug-resistant organisms (MDRO) via rectal swab at baseline (admission or within 14 days prior). MDROs include ESBL-producing Enterobacterales, carbapenem-resistant Enterobacterales (CRE), carbapenem-resistant Pseudomonas aeruginosa (CRPA), Acinetobacter baumannii (CRAB), and vancomycin-resistant Enterococcus (VRE).
Rate of Conversion from Negative to Positive MDRO Carriage During Hospitalization | From admission to discharge (up to 28 days)
  Proportion of participants who initially tested negative for MDRO digestive carriage at admission but later became positive on subsequent screening during hospitalization. Conversion will be assessed through weekly rectal swabs and swab at discharge.
Distribution of demographic and hospitalization-related characteristics among MDRO carriers | At enrollment
  Age, sex, and number of hospitalizations in the last 6 months among participants colonized with MDRO at enrollment
Prevalence of recent antibiotic use among MDRO carriers | At enrollment
  Proportion of MDRO carriers who received antibiotic treatment (at least 72 h) in the last 6 months, stratified by antibiotic class and duration
Charlson Comorbidity Index scores among MDRO carriers | At enrollment
  The Charlson Comorbidity Index (CCI) will be used to assess the burden of comorbidities at enrollment among participants with digestive MDRO carriage. The CCI score is calculated based on the presence of predefined conditions (e.g., diabetes, cancer, chronic heart failure), each assigned a weight, resulting in a total score ranging from 0 to 33.

CONTACTS AND LOCATIONS:
Locations (1):
- Emergency and Clinical Hospital Dr. Agrippa Ionescu, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to data protection regulations (GDPR - EU 2016/679) and the ethical requirement to ensure confidentiality of participant-level data. Only aggregated, anonymized results may be published.